CLINICAL TRIAL: NCT05212974
Title: COVID-19 Vaccine Hesitancy Among Nurses
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106114RINA
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Vaccine Hesitancy; Vaccination; Nurses
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses: Adult (≥ 20 and ≤80 years) male and female participants with verification of registered nurse license.
  Interventions: Other: Questionnaires
- General publics: Adult (≥ 20 and ≤80 years) male and female participants with reading abilities above the intermediate level.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The questionnaires include demographic data and vaccine hesitancy questions in a total of 35 items.

SUMMARY:
The purpose of this study is to investigate the correlation of intention to receive COVID-19 vaccine, recommendation behavior, and 5C psychological antecedents among Nurses. The results can be used to assist suggestions in the health education provided by nurses on the topic of COVID-19 pneumonia and its vaccination. The purpose of the study is also wants to build a basis for future research and public support in vaccine decision-making, as well as to enhance the promotion of vaccine policy and enhance the resilience of the whole population during the pandemic ear.

DETAILED DESCRIPTION:
A cross-sectional study based on convenience samples. The investigators recruit nurses and the general public to respond to structured self-filling electronic questionnaires by using an electronic data collection system. The questionnaires include demographic data and vaccine hesitancy questions in a total of 35 items. Convenience sampling was applied to estimate the sample size according to the number of nurses in each county. It is planned to collect a total of 4258 responses by the end of the study. The study instrument is the 5C psychological antecedents of vaccination, which includes Confidence, Complacency, Constraints, Calculation, and Collective Responsibility.

ELIGIBILITY:
[Nurses]

Inclusion Criteria:

* Male and female participants must be ≥ 20 years at the time of informed consent.
* Male and female participants have verification of registered nurse license.

Exclusion Criteria:

* Male and female participants be>80 years at the time of informed consent.

[General publics]

Inclusion Criteria:

* Male and female participants must be ≥ 20 years at the time of informed consent.
* Male and female participants have reading abilities above the intermediate level.

Exclusion Criteria:

* Male and female participants be>80 years at the time of informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: [Nurses] Adult (≥ 20 and ≤80 years) male and female participants with verification of registered nurse license.
  [General publics] Adult (≥ 20 and ≤80 years) male and female participants with reading abilities above the intermediate level.
Sampling Method: Non-Probability Sample
Enrollment: 4258 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
The correlation of intention to receive COVID-19 vaccine and 5C psychological antecedents (5C scale) among nurses and general publics. | The questionnaire length around 10 minutes.
  The 5C scale measures the psychological antecedents of vaccination, using 15 item tools including 5 domains (confidence, complacency, constraints, calculation, and collective responsibility). Each domain was assessed by 3 rating items on a 7-point scale (1=strongly disagree; 7=strongly agree). The mean scores of items under each domain were computed, with a higher average score indicating stronger agreement of the corresponding domain.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Chen Chang, Ph.D, Principal Investigator — Department of Nursing, National Taiwan University
Locations (1):
- Department of Nursing, National Taiwan University, Taipei, Taiwan